CLINICAL TRIAL: NCT03954210
Title: SIESTA: Sleep Intervention to Enhance Cognitive Status and Reduce Beta Amyloid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00143545; R01AG058530 (NIH)
Record Dates: First submitted 2019-05-13; First posted 2019-05-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Insomnia
Keywords: Cognitive Behavioral Therapy for Insomnia; CBT-I; Alzheimer's; Alzheimer's Disease
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Alzheimer Disease | interventions — Cognitive Behavioral Therapy; Sleep

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The research assistant will be blinded to the participant's intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Six-Week CBT-I Program (Experimental): CBT-I, six sessions, forty-five to sixty minutes in duration.
  Session 1: set up sleep restriction and stimulus control, discuss strategies for how to stay awake to a prescribed hour and what to do with wake after onset sleep time, provide sleep hygiene education.
  Session 2: determine if upward titration of total sleep time is warranted, review sleep hygiene.
  Session 3: continue upward titration of total sleep time, cognitive therapy for negative sleep beliefs if indicated.
  Session 4: continue upward titration of total sleep time, follow-up regarding negative sleep beliefs.
  Session 5: continue upward titration of total sleep time, discuss relapse prevention.
  Session 6: assess global treatment gains, discuss questions regarding relapse prevention.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)
- Six-Week Sleep and Lifestyle Education Program (Active Comparator): Sleep and Lifestyle Education, six sessions, forty-five to sixty minutes in duration.
  Session 1: Sleep education, Instruction/demonstration on stretching exercises.
  Session 2: Education on environmental factors & sleeping positions that impact sleep.
  Session 3: Education on lifestyle factors that impact sleep.
  Session 4: Education on diet and sleep.
  Session 5: Education on exercises and sleep.
  Session 6: Discus maintaining achievements & preventing relapses.
  Interventions: Behavioral: Sleep and Lifestyle Education

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — CBT-I is an in-person, one-on-one program with a graduate psychology research assistant who is trained in providing a standardized CBT-I. Participants will maintain a sleep diary during the course of the program to aid in tailoring the program. Each session will begin with a summary and graphing of sleep diary data and will include an assessment of treatment gains and adherence.
  Arms: Six-Week CBT-I Program
Behavioral: Sleep and Lifestyle Education — Participants in the sleep and lifestyle education group will attend six weekly, in-person, one-on-one, stretching, and thinking activity sessions with a graduate research assistant to control for socialization and contact with research personnel.
  Arms: Six-Week Sleep and Lifestyle Education Program

SUMMARY:
The objective of this study is to compare the efficacy of a sleep intervention on improving cognitive function in older adults with symptoms of insomnia, determine the association between change in sleep measures and change in cognitive function, and examine the efficacy of the sleep intervention on reducing the rate of Aβ deposition. Participants, ages 60-85, will be randomly assigned to a six-week sleep intervention program. A sub-group of fifty participants will undergo Florbetapir-Positron-emission tomography (PET) imaging during the one-year reassessment to examine the efficacy of the sleep intervention on reducing the rate of Aβ accumulation from baseline to one-year post-intervention.

DETAILED DESCRIPTION:
Lifestyle interventions to increase exercise and improve diet have been the focus of recent clinical trials to potentially prevent Alzheimer's disease (AD). However, despite the strong links between sleep disruptions, cognitive decline, and AD, sleep enhancement has yet to be targeted as a lifestyle intervention to prevent AD. Approximately fifteen percent of AD may be prevented by an efficacious intervention aimed to reduce sleep disturbances and sleep disorders. Chronic insomnia is the most frequent sleep disorder occurring in at least forty percent of older adults. Individuals with insomnia are more likely to be diagnosed with AD and demonstrate a decline in cognitive function at long-term follow-up. AD is characterized by the accumulation of Aβ plaques and tau tangles in the brain, and growing evidence shows impaired sleep contributes to the accumulation of Aβ. An intervention aimed at improving insomnia may represent a critical opportunity for primary prevention to slow cognitive decline and potentially delay the onset of AD. Therefore, the long-term goal of this research agenda is to understand how addressing sleep disturbances, via sleep intervention, may delay the onset of AD.

ELIGIBILITY:
Inclusion Criteria:

* Report of difficulty falling asleep, maintaining sleep, or waking up too early at least three nights a week for the past six months
* A score of greater than, or equal to, ten on the Insomnia Severity Index
* A score of greater than, or equal to, twenty-five on the Mini-Mental State Examination (MMSE)
* A score of less than, or equal to, two on the Dementia Screening Interview (AD8)

Exclusion Criteria:

* A known untreated sleep disorder (i.e., sleep apnea or restless leg syndrome)
* Currently taking benzodiazepines, non-benzodiazepines, melatonin supplements, or agonists for insomnia
* A score of greater than, or equal to, fifteen on the Patient Health Questionnaire (PHQ-9) indicating severe depression or endorsement of any suicidal ideation (an answer of one, two, or three on item number nine of the PHQ-9)
* History of drug or alcohol abuse as defined by the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-4) criteria within the last two years
* History of a nervous system disorder (i.e., stroke, Parkinson's Disease)
* Severe mental illness (i.e., Schizophrenia, Bipolar Disorder)
* History of a learning disability or attention-deficit/hyperactivity disorder
* Current, or history of, shift work
* Currently receiving CBT-I treatment
* Unable to hear at a conversational level
* Failure of a near vision test utilizing the Logarithmic Near Visual Acuity Chart

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Continuous Performance Test (CPT) | Baseline, 6-Week Reassessment, and One-Year Reassessment
  Assessment of the participants attention. Participants will be given a set of rules for stimuli, and based on those rules they will determine if a presented stimuli fit within those rules. Scores will be determined by the number of correctly identified stimuli.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Baseline, 6-Week Reassessment, and One-Year Reassessment
  Twelve sub-tests assessing participants immediate memory, visuospatial/constructional, language, attention, and delayed memory skills.Participants will engage in list learning, story memory, figure copying, line orientation, picture naming, semantic fluency, digit span, coding, list recall, list recognition, story memory and figure recall.
Stroop Test | Baseline, 6-Week Reassessment, and One-Year Reassessment
  Assessment of participants executive functioning. Participants will be required to inhibit their natural response and replace it with a different response (i.e., reading a word versus saying the color of the word). Scores are obtained by taking the difference between conditions and normalizing for the number of stimuli.
Neuropsychological Assessment Battery-Digits Forward/Digits Backward Test | Baseline, 6-Week Reassessment, and One-Year Reassessment
  Assessment of the participants attention and working memory. Participants will be required to remember and recall strings of numbers ranging from three to nine. Primary scores are obtained by tallying the number of trials the participant accurately recalled in the forward direction and the backward direction. Secondary scores are obtained by determining the longest string of numbers the participant recalled in the forward and backward direction.

SECONDARY OUTCOMES:
Polysomnography | Second Pre-Screening/Baseline, 6-Week Reassessment, and One-Year Assessment
  Assessment to determine if the participants have a sleep disorder. This determination is made by a trained professional utilizing the patient's brain waves, blood oxygen level, heart rate, breathing, and eye and leg movements to determine.

OTHER OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Pre-Screening/Baseline, 6-Week Reassessment and One-Year Reassessment
  Assessment of patients depression over the past two weeks. There are nine items that yield a maximum score of twenty-seven. Each item is anchored on a four-point scale with 0 being "Not at all" and 3 being "Nearly Everyday." Participants can demonstrate a minimum score of zero (no depression) or twenty-seven (severe depression). The tenth item that assesses how depressive symptoms affect functional level will not be utilized.
Generalized Anxiety Disorder Assessment (GAD-7) | Baseline, 6-Week Reassessment, and One-Year Reassessment
  Assessment of patients anxiety over the past two weeks. There are eight items anchored on a scale of zero ("Not at all") to three ("Nearly Everyday"), that yield a minimum score of zero (no anxiety) and a maximum score of twenty-one (daily anxiety). An additional item was added to assess if anxiety impacts daily activities and sociability.
Sleep Efficacy Scale (SES) | Baseline, 6-Week Reassessment, and One-Year Reassessment
  Assessment of patients level of confidence in being able to implement behaviors that are helpful in promoting sleep. There are nine items that are scored on a four-point scale ranging from one (not confident) to five (very confident), with a minimum score of nine, indicating lower self-efficacy, and a maximum score of forty-five indicating higher self-efficacy.
Florbetapir PET Imaging | Baseline and One-Year Assessment
  2D imaging technique utilized to assess change in Beta Amyloid deposition in the brain over time.Interested brain areas include the frontal lobes, anterior cingulate, posterior cingulate, parietal lobes and temporal lobes.
Magnetic Resonance Imaging (MRI) | Baseline and One-Year Assessment
  3D imaging technique utilized to assess change in Beta Amyloid deposition in the brain over time. Interested brain areas include the frontal lobes, anterior cingulate, posterior cingulate, parietal lobes and temporal lobes.
Motivation to Change Sleep Behaviors | Baseline
  Participants self-reported desire to change their current sleep behaviors. Participants will answer one item based on a five-point Likert scale ranging from zero (not at all motivated) to four (very motivated). A minimum score of zero can be obtained indicating no motivation to change sleep behaviors and a maximum score of five indicating high motivation to change sleep behaviors.
Mini Mental-State Examination (MMSE) | Second Pre-Screening
  Assessment of mild cognitive impairment. Participants are required to answer, or complete, eleven items. For this study, participants with a score of greater than, or equal to twenty-five will be considered mildly cognitively impaired and will be excluded from the study.
Logarithmic Near Visual Acuity Chart | Second Pre-Screening
  Assessment of near visual acuity based on a standardized vision chart placed sixteen inches away from the participant's eyes.
Apolipoprotein E (APOE) 4 Genotyping | Baseline
  A blood draw of twenty milliliters utilized to determine if a participant may have probable late onset Alzheimer's disease.
Coin in Hand | Baseline, 6-Week Reassessment, and One-Year Reassessment
  Assessment of the participants effort to ensure full effort is being given during testing.
Grooved Pegboard Test | Baseline, 6-Week Reassessment, and One-Year Reassessment
  Assessment of the participants speed at completing a task requiring fine motor skills. Outcome is the amount of time required for the participant to place twenty-five pegs into the pegboard first utilizing their dominant hand only, then using their non-dominant hand only.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Siengsukon, PT, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center- Sleep, Health and Wellness Laboratory, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available to other researchers. However, the results of this study will be registered to ClinicalTrials.gov within twelve months of the primary study completion date including information about participant flow, demographic and baseline characteristics, outcomes and statistical analyses, adverse events, the protocol, and statistical analysis plan, and administrative information. In addition, results will be disseminated via oral presentations and news stories in collaboration with the University of Kansas Medical Center public relations team and local news outlets.

REFERENCES:
- [Background] Solomon A, Mangialasche F, Richard E, Andrieu S, Bennett DA, Breteler M, Fratiglioni L, Hooshmand B, Khachaturian AS, Schneider LS, Skoog I, Kivipelto M. Advances in the prevention of Alzheimer's disease and dementia. J Intern Med. 2014 Mar;275(3):229-50. doi: 10.1111/joim.12178. PMID 24605807
- [Background] Wang J, Tan L, Yu JT. Prevention Trials in Alzheimer's Disease: Current Status and Future Perspectives. J Alzheimers Dis. 2016;50(4):927-45. doi: 10.3233/JAD-150826. PMID 26836177
- [Background] Bubu OM, Brannick M, Mortimer J, Umasabor-Bubu O, Sebastiao YV, Wen Y, Schwartz S, Borenstein AR, Wu Y, Morgan D, Anderson WM. Sleep, Cognitive impairment, and Alzheimer's disease: A Systematic Review and Meta-Analysis. Sleep. 2017 Jan 1;40(1). doi: 10.1093/sleep/zsw032. PMID 28364458
- [Background] Alessi C, Vitiello MV. Insomnia (primary) in older people: non-drug treatments. BMJ Clin Evid. 2015 May 13;2015:2302. PMID 25968443
- [Background] Lobo A, Lopez-Anton R, de-la-Camara C, Quintanilla MA, Campayo A, Saz P; ZARADEMP Workgroup. Non-cognitive psychopathological symptoms associated with incident mild cognitive impairment and dementia, Alzheimer's type. Neurotox Res. 2008 Oct;14(2-3):263-72. doi: 10.1007/BF03033815. PMID 19073431
- [Background] Osorio RS, Pirraglia E, Aguera-Ortiz LF, During EH, Sacks H, Ayappa I, Walsleben J, Mooney A, Hussain A, Glodzik L, Frangione B, Martinez-Martin P, de Leon MJ. Greater risk of Alzheimer's disease in older adults with insomnia. J Am Geriatr Soc. 2011 Mar;59(3):559-62. doi: 10.1111/j.1532-5415.2010.03288.x. No abstract available. PMID 21391952
- [Background] Cricco M, Simonsick EM, Foley DJ. The impact of insomnia on cognitive functioning in older adults. J Am Geriatr Soc. 2001 Sep;49(9):1185-9. doi: 10.1046/j.1532-5415.2001.49235.x. PMID 11559377
- [Background] Ju YE, Lucey BP, Holtzman DM. Sleep and Alzheimer disease pathology--a bidirectional relationship. Nat Rev Neurol. 2014 Feb;10(2):115-9. doi: 10.1038/nrneurol.2013.269. Epub 2013 Dec 24. PMID 24366271
- [Background] Branger P, Arenaza-Urquijo EM, Tomadesso C, Mezenge F, Andre C, de Flores R, Mutlu J, de La Sayette V, Eustache F, Chetelat G, Rauchs G. Relationships between sleep quality and brain volume, metabolism, and amyloid deposition in late adulthood. Neurobiol Aging. 2016 May;41:107-114. doi: 10.1016/j.neurobiolaging.2016.02.009. Epub 2016 Feb 17. PMID 27103523
- [Background] Xie L, Kang H, Xu Q, Chen MJ, Liao Y, Thiyagarajan M, O'Donnell J, Christensen DJ, Nicholson C, Iliff JJ, Takano T, Deane R, Nedergaard M. Sleep drives metabolite clearance from the adult brain. Science. 2013 Oct 18;342(6156):373-7. doi: 10.1126/science.1241224. PMID 24136970
- [Background] Wang MY, Wang SY, Tsai PS. Cognitive behavioural therapy for primary insomnia: a systematic review. J Adv Nurs. 2005 Jun;50(5):553-64. doi: 10.1111/j.1365-2648.2005.03433.x. PMID 15882372
- [Background] Geiger-Brown JM, Rogers VE, Liu W, Ludeman EM, Downton KD, Diaz-Abad M. Cognitive behavioral therapy in persons with comorbid insomnia: A meta-analysis. Sleep Med Rev. 2015 Oct;23:54-67. doi: 10.1016/j.smrv.2014.11.007. Epub 2014 Nov 29. PMID 25645130
- [Background] Trauer JM, Qian MY, Doyle JS, Rajaratnam SM, Cunnington D. Cognitive Behavioral Therapy for Chronic Insomnia: A Systematic Review and Meta-analysis. Ann Intern Med. 2015 Aug 4;163(3):191-204. doi: 10.7326/M14-2841. PMID 26054060
- [Background] Wu JQ, Appleman ER, Salazar RD, Ong JC. Cognitive Behavioral Therapy for Insomnia Comorbid With Psychiatric and Medical Conditions: A Meta-analysis. JAMA Intern Med. 2015 Sep;175(9):1461-72. doi: 10.1001/jamainternmed.2015.3006. PMID 26147487
- [Background] Diekelmann S, Wilhelm I, Born J. The whats and whens of sleep-dependent memory consolidation. Sleep Med Rev. 2009 Oct;13(5):309-21. doi: 10.1016/j.smrv.2008.08.002. Epub 2009 Feb 28. PMID 19251443
- [Background] CDC. Insufficient sleep is a public health problem. http://www.cdc.gov/features/dssleep/. Accessed 1/29/16.
- [Background] Hahn EA, Wang HX, Andel R, Fratiglioni L. A change in sleep pattern may predict Alzheimer disease. Am J Geriatr Psychiatry. 2014 Nov;22(11):1262-71. doi: 10.1016/j.jagp.2013.04.015. Epub 2013 Aug 14. PMID 23954041
- [Background] Lim AS, Kowgier M, Yu L, Buchman AS, Bennett DA. Sleep Fragmentation and the Risk of Incident Alzheimer's Disease and Cognitive Decline in Older Persons. Sleep. 2013 Jul 1;36(7):1027-1032. doi: 10.5665/sleep.2802. PMID 23814339
- [Background] Ju YE, McLeland JS, Toedebusch CD, Xiong C, Fagan AM, Duntley SP, Morris JC, Holtzman DM. Sleep quality and preclinical Alzheimer disease. JAMA Neurol. 2013 May;70(5):587-93. doi: 10.1001/jamaneurol.2013.2334. PMID 23479184
- [Background] Bero AW, Yan P, Roh JH, Cirrito JR, Stewart FR, Raichle ME, Lee JM, Holtzman DM. Neuronal activity regulates the regional vulnerability to amyloid-beta deposition. Nat Neurosci. 2011 Jun;14(6):750-6. doi: 10.1038/nn.2801. Epub 2011 May 1. PMID 21532579
- [Background] Varga AW, Wohlleber ME, Gimenez S, Romero S, Alonso JF, Ducca EL, Kam K, Lewis C, Tanzi EB, Tweardy S, Kishi A, Parekh A, Fischer E, Gumb T, Alcolea D, Fortea J, Lleo A, Blennow K, Zetterberg H, Mosconi L, Glodzik L, Pirraglia E, Burschtin OE, de Leon MJ, Rapoport DM, Lu SE, Ayappa I, Osorio RS. Reduced Slow-Wave Sleep Is Associated with High Cerebrospinal Fluid Abeta42 Levels in Cognitively Normal Elderly. Sleep. 2016 Nov 1;39(11):2041-2048. doi: 10.5665/sleep.6240. PMID 27568802
- [Background] Ohayon MM, Carskadon MA, Guilleminault C, Vitiello MV. Meta-analysis of quantitative sleep parameters from childhood to old age in healthy individuals: developing normative sleep values across the human lifespan. Sleep. 2004 Nov 1;27(7):1255-73. doi: 10.1093/sleep/27.7.1255. PMID 15586779
- [Background] Merica H, Blois R, Gaillard JM. Spectral characteristics of sleep EEG in chronic insomnia. Eur J Neurosci. 1998 May;10(5):1826-34. doi: 10.1046/j.1460-9568.1998.00189.x. PMID 9751153
- [Background] Pigeon WR, Perlis ML. Sleep homeostasis in primary insomnia. Sleep Med Rev. 2006 Aug;10(4):247-54. doi: 10.1016/j.smrv.2005.09.002. Epub 2006 Mar 24. PMID 16563817
- [Background] Cervena K, Dauvilliers Y, Espa F, Touchon J, Matousek M, Billiard M, Besset A. Effect of cognitive behavioural therapy for insomnia on sleep architecture and sleep EEG power spectra in psychophysiological insomnia. J Sleep Res. 2004 Dec;13(4):385-93. doi: 10.1111/j.1365-2869.2004.00431.x. PMID 15560773
- [Background] Foley D, Monjan A, Masaki K, Ross W, Havlik R, White L, Launer L. Daytime sleepiness is associated with 3-year incident dementia and cognitive decline in older Japanese-American men. J Am Geriatr Soc. 2001 Dec;49(12):1628-32. doi: 10.1046/j.1532-5415.2001.t01-1-49271.x. PMID 11843995
- [Background] Kreutzmann JC, Havekes R, Abel T, Meerlo P. Sleep deprivation and hippocampal vulnerability: changes in neuronal plasticity, neurogenesis and cognitive function. Neuroscience. 2015 Nov 19;309:173-90. doi: 10.1016/j.neuroscience.2015.04.053. Epub 2015 Apr 29. PMID 25937398
- [Background] Mitchell MD, Gehrman P, Perlis M, Umscheid CA. Comparative effectiveness of cognitive behavioral therapy for insomnia: a systematic review. BMC Fam Pract. 2012 May 25;13:40. doi: 10.1186/1471-2296-13-40. PMID 22631616
- [Background] Musiek ES, Xiong DD, Holtzman DM. Sleep, circadian rhythms, and the pathogenesis of Alzheimer disease. Exp Mol Med. 2015 Mar 13;47(3):e148. doi: 10.1038/emm.2014.121. PMID 25766617
- [Background] Vitiello MV, McCurry SM, Shortreed SM, Balderson BH, Baker LD, Keefe FJ, Rybarczyk BD, Von Korff M. Cognitive-behavioral treatment for comorbid insomnia and osteoarthritis pain in primary care: the lifestyles randomized controlled trial. J Am Geriatr Soc. 2013 Jun;61(6):947-956. doi: 10.1111/jgs.12275. Epub 2013 May 27. PMID 23711168
- [Background] McCurry SM, Shortreed SM, Von Korff M, Balderson BH, Baker LD, Rybarczyk BD, Vitiello MV. Who benefits from CBT for insomnia in primary care? Important patient selection and trial design lessons from longitudinal results of the Lifestyles trial. Sleep. 2014 Feb 1;37(2):299-308. doi: 10.5665/sleep.3402. PMID 24497658
- [Derived] Hand LK, Key MN, Vidoni ED, Ludwig R, Nelson E, Glaser A, Drerup M, Phadnis MA, Bruce J, Burns JM, Siengsukon CF. Sleep Fragmentation and Sleep Stages 1 and 2 Are Associated With Amyloid-Beta Burden in Cognitively Normal Older Adults. J Sleep Res. 2025 Jun 3:e70098. doi: 10.1111/jsr.70098. Online ahead of print. PMID 40461009